CLINICAL TRIAL: NCT05499676
Title: Development and Pilot Testing of a Cognitive-Behavioral Therapy-Guided Self-Help Mobile App for the Post-Acute Treatment of Anorexia Nervosa
Brief Title: Helping HAND: Healing Anorexia Nervosa Digitally
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ellen E. Fitzsimmons-Craft, Associate Professor of Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202202113; R34MH127203 (NIH)
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mobile Coached Intervention (Experimental): Participants randomized to the mobile intervention condition will receive access to the mobile app for 6 consecutive months. Participants will still be able to access other usual care options and will be encouraged to follow the discharge plan provided to them by the eating disorder program from which they were discharged.
  Interventions: Device: SilverCloud Health Mobile Intervention
- Mobile Coached Intervention Plus Social Networking (Experimental): Participants randomized to the mobile intervention plus social networking condition will receive access to the mobile app, as well as Facebook social networking component, for 6 consecutive months. Participants will still be able to access other usual care options and will be encouraged to follow the discharge plan provided to them by the eating disorder program from which they were discharged.
  Interventions: Device: SilverCloud Health Mobile Intervention; Device: Social Networking Intervention: Facebook
- Treatment as Usual (No Intervention): This group will be encouraged to follow the discharge plan provided to them by the eating disorder program from which they were discharged. Participants will also be encouraged to follow-up with their eating program for additional referral information as needed and/or to reach out to the National Eating Disorders Association (NEDA) and/or Association for Anorexia Nervosa and Associated Disorders (ANAD ) for assistance with finding treatment providers/resources as needed. NEDA and ANAD provide helplines and online treatment provider databases to help individuals find providers.

INTERVENTIONS:
Device: SilverCloud Health Mobile Intervention — SilverCloud Health is a mobile mental health platform offering cognitive-behavioral therapy-based guided self-help programs, including one for anorexia nervosa developed by our team. Participants in this arm will receive the support of a coach to guide them through the program. Participants will be able to communicate with their coach within the program.
  Arms: Mobile Coached Intervention; Mobile Coached Intervention Plus Social Networking
Device: Social Networking Intervention: Facebook — Facebook is a social networking site that will offer participants the opportunity to interact with study team posts, post themselves, and connect with others in the study experiencing similar struggles in a private group
  Arms: Mobile Coached Intervention Plus Social Networking

SUMMARY:
The proposed project will develop and pilot a coached mobile app, including a social networking component, for individuals with anorexia nervosa to use in the post-acute period

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a costly and life-threatening illness. Patients with severe AN are often treated in the acute setting, but relapse after treatment is common. Further, the discharge criterion in acute settings is typically weight restoration. However, research has indicated that weight-based recovery is not "enough" and that full recovery involves physical, behavioral, and psychological components. Cognitive-behavioral therapy (CBT) is useful with this population, including following discharge, and may aid in addressing psychological symptoms, achieving full recovery, and decreasing relapse. However, very few patients have access to providers trained in these techniques. mHealth technologies have great potential to exponentially increase access to high-quality services for the post-acute treatment of AN by addressing barriers to treatment, but to date, research on these approaches has been extremely limited. A guided self-help CBT-based mobile app, StudentBodies-Eating Disorders (SB-ED), has been successfully developed, demonstrating effectiveness among college women with binge/purge-type EDs. At the same time, there is demonstrated support for in-person CBT for the post-acute care and relapse prevention of adult AN. The overarching goal of this R34 is thus to develop and test a CBT-based, coached mobile app to address the post-acute care and relapse prevention.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender women who are 18 years old and older, who own a mobile phone, speak English, are U.S. residents, have a BMI greater than or equal to 17, who are connected with a physician (such as a primary care provider), who are not using a feeding tube, and who have been discharged from intensive treatment (i.e., inpatient, residential, partial hospitalization, intensive outpatient) for DSM-5 anorexia nervosa within the past 2 months.

Exclusion Criteria:

* Individuals who are not cisgender women.
* Individuals under 18 years old.
* Individuals who do not own a mobile phone.
* Individuals who have not been discharged from intensive treatment (i.e., inpatient, residential, partial hospitalization, intensive outpatient) for DSM-5 anorexia nervosa within the past 2 months).
* Individuals who are not connected with a physician (such as a primary care provider)
* Individuals who have a BMI below 17.0
* Individuals who are currently using a feeding tube

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender women
Enrollment: 90 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
1. Effectiveness of the mobile app conditions, compared to referral to usual care, in changing eating disorder psychopathology, as assessed by the Eating Disorder Examination-Questionnaire. | baseline, 6 months, and 9 months
  Investigators will use the Eating Disorder Examination-Questionnaire (EDE-Q), a 28-item measure derived from a diagnostic interview, the standard measure of eating disorder psychopathology. The main outcome variable will be the EDE-Q Global score, an overall measure of eating disorder psychopathology. Scores possible range from 0 to 6, with higher scores indicating greater eating disorder psychopathology. Change in EDE-Q scores will be compared from baseline to 6 months and baseline to 9 months.

SECONDARY OUTCOMES:
Effectiveness of the mobile app conditions, compared to referral to usual care, in changing eating disorder behaviors. | baseline, 6 months, and 9 months
  Investigators will use the Eating Disorder Examination-Questionnaire (EDE-Q), a 28-item measure derived from a diagnostic interview, the standard measure of eating disorder psychopathology. For this secondary outcome, investigators will examine eating disorder behavior frequencies from the EDE-Q. Change in EDE-Q behavior frequencies will be compared from baseline to 6 months and baseline to 9 months.
Effectiveness of the mobile app conditions, compared to referral to usual care, in changing Body Mass Index (BMI). | baseline, 6 months, and 9 months
  Investigators will use current BMI as derived from self-reported height, which has shown to be accurate in adult ED populations, and weight assessed by a digital wireless scale. At each of the study timepoints, a study coordinator will schedule a time with the participant to take their weight while they are on a Zoom call with the coordinator.
  Participants will be instructed to take off their shoes, wear light clothing, and empty their pockets, similar to the instructions that would be provided if this measurement were being taken in person. Given the use of a wireless scale, the measurement will be able to be immediately and automatically sent to the research team. Change in BMI will be compared from baseline to 6 months and baseline to 9 months.
Effectiveness of the mobile app conditions, compared to referral to usual care, in changing depression and suicidal ideation, as assessed by the Patient Health Questionnaire. | baseline, 6 months, and 9 months
  Investigators will use the Patient Health Questionnaire (PHQ-9), a 9-item measure that is widely used to assess presence of possible depression and severity, as well as suicidality. Scores possible range from 0 to 27, with higher scores indicating greater severity of depression. Change in PHQ scores will be compared from baseline to 6 months and baseline to 9 months.
Effectiveness of the mobile app conditions, compared to referral to usual care, in changing clinical impairment, as assessed by the Clinical Impairment Assessment. | baseline, 6 months, and 9 months
  Investigators will use the Clinical Impairment Assessment (CIA), which is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features. Scores range from 0 to 48 with higher scores indicating higher levels of impairment. Change in CIA scores will be compared from baseline to 6 months and baseline to 9 months.

OTHER OUTCOMES:
Effectiveness of the mobile app conditions, compared to referral to usual care, in terms of reducing rehospitalization. | 6 months and 9 months
  To assess rehospitalization and other treatment utilization, investigators will use a detailed treatment history questionnaire. Rehospitalization rates will be compared across conditions at 6 months and 9 months.
Effectiveness of the mobile app conditions, compared to referral to usual care, in terms of achieving full recovery, as assessed with BMI, the Stanford-Washington University Eating Disorders Screen, and the EDE-Q. | 6 months and 9 months
  For recovery, at 6- and 9-month assessments, investigators will compare the percent of participants across study conditions who have achieved full recovery from an eating disorder, comprised of: 1) physical recovery based on having a BMI ≥ 18.5 kg/m2; 2) behavioral recovery based on absence of binge eating, vomiting, laxative use, and fasting in the past 3 months (assessed via the Stanford-Washington University Eating Disorder Screen); and 3) cognitive recovery based on scoring within 1 SD of community norms for each of the EDE-Q subscales.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Palo Alto University, Palo Alto, California
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: No
De-identified data will not be shared on the National Institute of Mental Health Data Archive, as this is a pilot study.